CLINICAL TRIAL: NCT00421889
Title: A Phase I/II Safety, Pharmacodynamic, and Pharmacokinetic Study of Intravenously Administered PXD101 Plus Carboplatin or Paclitaxel or Both in Patients With Advanced Solid Tumours
Brief Title: A Study of Belinostat + Carboplatin or Paclitaxel or Both in Patients With Ovarian Cancer in Need of Relapse Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PXD101-CLN-8; PXD101-040-EU
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Ovarian Cancer; Epithelial Ovarian Cancer; Fallopian Tube Cancer; Bladder Cancer
Keywords: Ovarian cancer; Ovarian Neoplasms; Primary peritoneal; Epithelial ovarian; Fallopian tube; Bladder cancer; belinostat; PXD101; mixed mullerian cancer of ovarian origin
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Urinary Bladder Neoplasms | interventions — belinostat; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Belinostat: 1000 mg/m2 days 1-5 in a 21 day cycle; IV Paclitaxel: Administered IV 2-3 hours after belinostat infusion on day 3 in a 21-day cycle
  Carboplatin: Administered IV infusion after paclitaxel on day 3 in a 21-day cycle
  Interventions: Drug: belinostat; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: belinostat
  Other Names: PXD101
Drug: Paclitaxel
Drug: Carboplatin

SUMMARY:
The study seeks to assess the safety, pharmacodynamics, pharmacokinetics and efficacy of belinostat (PXD101) administered in combination with carboplatin or paclitaxel or both in patients with solid tumours followed by maximum tolerated dose (MTD) expansion (phase II) in ovarian and bladder cancer patients

The clinical trial is now in the MTD (phase II) portion of the study enrolling bladder cancer patients. Enrollment of ovarian patients is complete.

DETAILED DESCRIPTION:
MTD Expansion I(Phase II): A total of 18-32 patients with epithelial ovarian, primary peritoneal, fallopian tube or mixed mullerian tumours of ovarian origin, in need of relapse treatment will be enrolled.

MTD Expansion II (phase II): A total of 15 patients with urothelial (transitional cell) carcinoma of the bladder will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent of an IRB (Institutional Review Board) approved consent form.
2. Patients with histologically confirmed solid carcinomas, for which there is no known curative therapy.
3. Performance status (Eastern Cooperative Oncology Group [ECOG]) ≤ 2.
4. Life expectancy of at least 3 months.
5. Age ≥ 18 years.
6. Acceptable liver, renal and bone marrow function including the following:

   1. Bilirubin ≤ 1.5 times ULN (upper limit of normal).
   2. AST/SGOT ([Aspartate Amino Transferase/Serum glutamic oxaloacetic transaminase]), ALT/SGPT ([Alanine Amino Transferase/Serum glutamic pyruvic transaminase]) and alkaline phosphatase ≤ 3 times ULN (if liver metastases are present, then ≤ 5 x ULN is allowed).
   3. Measured EDTA ([ethylenediaminetetraacetic acid]) renal clearance ≥ 45 mL/min (EU sites). At the US sites calculated creatinine clearance ≥ 45 mL/min using the Jeliffe formula.
   4. Leukocytes > 2.5×109/L, neutrophils > 1.0x109/L, platelets > 100×109/L.
   5. Hemoglobin > 9.0 g/dL or > 5.6 mmol/L.
7. Acceptable coagulation status: PT-INR([prothrombin-International Normalized Ratio])/APTT([Activated Partial Thromboplastin Time]) ≤ 1.5 × ULN or in the therapeutic range if on anticoagulation therapy
8. A negative pregnancy test for women of childbearing potential. For men and women of child-producing potential, the use of effective contraceptive methods during the study is required.
9. Serum potassium within normal range (added in protocol Global version 3.0) Additional Eligibility Criteria at the MTD Expansion only
10. Patients with epithelial ovarian cancer in need of relapse treatment. Changed with protocol Global version 3 to: Patients with epithelial ovarian, primary peritoneal, fallopian tube or mixed mullerian tumors of ovarian origin in need of relapse treatment.

    Or
11. Patients with urothelial (transitional cell) carcinoma of the bladder who have received up to a maximum of 3 previous chemotherapy regimens in the advanced disease setting (neoadjuvant chemotherapy is not included in the total of chemotherapy regimens), applies only for patients enrolled in Part D.
12. At least one uni-dimensional measurable lesion. Lesions must be measured by CT scan or MRI according to Response Evaluation Criteria in Solid Tumors (RECIST)(Added with protocol Global version 4).

    Eligibility Criteria for the Site Specific Amendment (Part C) - Advanced solid tumors only
13. Patients with refractory solid tumors other than ovarian cancer.

Exclusion Criteria:

1. Treatment with investigational agents within the last 4 weeks.
2. Prior anticancer therapy within the last 3 weeks of study dosing including chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of other investigational agents. Changed with protocol Global version 1; prior anticancer therapy within the last 3 weeks of study dosing including chemotherapy, radiotherapy, endocrine therapy or immunotherapy.
3. Co-existing active infection or any co-existing medical condition likely to interfere with study procedures, including significant cardiovascular disease (New York Heart Association Class III or IV cardiac disease), myocardial infarction within the past 6 months, unstable angina, congestive heart failure requiring therapy, unstable arrhythmia or a need for anti-arrhythmic therapy, or evidence of ischemia on ECG, marked baseline prolongation of QT/QTc interval, e.g., repeated demonstration of a QTc interval ([corrected QT interval ]) > 500 msec; Long QT Syndrome; the required use of concomitant medication on belinostat infusion days that may cause Torsade de Pointes (see Appendix 1.1, protocol EU version 1.0, Appendix A - Appendix 16.1.1).
4. Altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies.
5. History of a concurrent second malignancy. Changed with Site Specific Amendment (Part D) to: History of a concurrent second malignancy. In patients with urothelial (transitional cell) carcinoma of the bladder an exception is that an incidental finding of localized prostate cancer at the time of radical cystectomy does not preclude inclusion in the study. In such cases a patient will be eligible for inclusion if the Gleason score is ≤6 and the Prostate Specific Antigen (PSA) <10 ng/mL (if the patient would be on hormonal treatment the PSA must be undetectable).Only applied to patients included in this site specific amendment.
6. History of hypersensitivity to either platinum or paclitaxel that is unable to be desensitized (added with protocol Global version 4).
7. More than 3 prior lines of chemotherapy given for metastatic disease (added with protocol Global version 1).
8. Bowel obstruction or impending bowel obstruction.
9. Known HIV positivity.
10. Any Grade 2 or above drug-related neurotoxicity, following recovery.
11. Changed with protocol Global version 1 to: Any existing Grade 2 or above drug related neurotoxicity due to prior treatment with agents causing neurotoxicity.

    Additional exclusion criteria at the MTD expansion only
12. Mixed mullerian tumors of intra-uterine origin, added with protocol Global version 3.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: e-mail contact via enquires@topotarget.com, Study Director — Valerio Therapeutics
Locations (11):
- United States (7):
  - Gynecologic Oncology Associates, Newport Beach, California
  - Research Facility, Orlando, Florida
  - Hematology and Oncology Specialists, LLC, Covington, Louisiana
  - Hematology & Oncology Specialists, LLC, Metairie, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
- Denmark (2):
  - The Finsen Center, Rigshospitalet, Copenhagen
  - Research Facility, Herlev University Hospital, Herlev
- United Kingdom (2):
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - The Royal Marsden NHS Trust, Surrey

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Dose Escalation 600/5/NA: PXD101: 600 mg/m2 30-minute IV infusion every 24 hours for 5 days every 3 weeks (period of 3 weeks is one cycle) Carboplatin: AUC 5 (area under the curve) administered 2-3 hours after PXD101 on Cycle Day 3 Paclitaxel: 0 mg/m2 administered 2-3 hours after PXD101 on Cycle Day 3
- Part A: Dose Escalation 600/NA/175: PXD101: 600 mg/m2 30-minute IV infusion every 24 hours for 5 days every 3 weeks (period of 3 weeks is one cycle) Carboplatin: None administered 2-3 hours after PXD101 on Cycle Day 3 Paclitaxel: 175 mg/m2 administered 2-3 hours after PXD101 on Cycle Day 3
- Part A: Dose Escalation 600/5/175: PXD101: 600 mg/m2 30-minute IV infusion every 24 hours for 5 days every 3 weeks (period of 3 weeks is one cycle) Carboplatin: AUC 5 administered 2-3 hours after PXD101 on Cycle Day 3 Paclitaxel: 175 mg/m2 administered 2-3 hours after PXD101 on Cycle Day 3
- Part A: Dose Escalation 800/5/175: PXD101: 800 mg/m2 30-minute IV infusion every 24 hours for 5 days every 3 weeks (period of 3 weeks is one cycle) Carboplatin: AUC 5 administered 2-3 hours after PXD101 on Cycle Day 3 Paclitaxel: 175 mg/m2 administered 2-3 hours after PXD101 on Cycle Day 3
- Part A: Dose Escalation 1000/5/175; Part B: Ovarian Cancer MTD: PXD101: 1000 mg/m2 30-minute IV infusion every 24 hours for 5 days every 3 weeks (period of 3 weeks is one cycle) Carboplatin: AUC 5 administered 2-3 hours after PXD101 on Cycle Day 3 Paclitaxel: 175 mg/m2 administered 2-3 hours after PXD101 on Cycle Day 3
- Part C: 3 Hours Infusion, Solid Tumors Except Ovarian Cancer: PXD: 1000 mg/m² was administered as a 3 hour IV infusion every 24 hours for 5 days on Day 1-5 every 3 weeks Paclitaxel: 175 mg/m² IV administered 2-3 hours following the infusion of PXD101 on cycle Day 3 Carboplatin: AUC of 5 IV administered 2-3 hours following the infusion of PXD101 on cycle Day 3 (carboplatin after paclitaxel)
- Part C: 6 Hours Infusion Solid Tumors, Except Ovarian Cancer: PXD: 1000 mg/m² was administered as a 6-hour IV infusion every 24 hours for 5 days on Day 1-5 every 3 weeks Paclitaxel: 175 mg/m² IV administered 2-3 hours following the infusion of PXD101 on cycle Day 3 Carboplatin: AUC of 5 IV administered 2-3 hours following the infusion of PXD101 on cycle Day 3 (carboplatin after paclitaxel)
- Part D: Bladder Cancer MTD: PXD101: 1000 mg/m² 30-minute IV infusion every 24 hours for 5 days on Day 1-5 every 3 weeks Carboplatin: AUC 5 IV, 2-3 hours following the infusion of PXD101 on Cycle Day 3 Paclitaxel: 175 mg/m² IV, 2-3 hours following the infusion of PXD101 on Cycle Day 3
Period: Overall Study
Arm/Group | Part A: Dose Escalation 600/5/NA | Part A: Dose Escalation 600/NA/175 | Part A: Dose Escalation 600/5/175 | Part A: Dose Escalation 800/5/175 | Part A: Dose Escalation 1000/5/175 | Part B: Ovarian Cancer MTD | Part C: 3 Hours Infusion, Solid Tumors Except Ovarian Cancer | Part C: 6 Hours Infusion Solid Tumors, Except Ovarian Cancer | Part D: Bladder Cancer MTD
Started | 5 | 5 | 3 | 4 | 6 | 35 | 4 | 3 | 15
Completed | 0 (Mean number of PXD101 cycles administered: 5.20) | 0 (Mean number of PXD101 cycles administered: 8.20) | 0 (Mean number of PXD101 cycles administered: 3.33) | 0 (Mean number of PXD101 cycles administered: 9.25) | 0 (Mean number of PXD101 cycles administered: 5.00) | 0 (Mean number of PXD101 cycles administered: 7.69) | 0 (Mean number of PXD101 cycles administered: 5.50) | 1 (Mean number of PXD101 cycles administered: 3.33) | 4 (Mean number of PXD101 cycles administered: 4.27)
Not Completed | 5 | 5 | 3 | 4 | 6 | 35 | 4 | 2 | 11
Not completed — Adverse Event | 1 | 0 | 1 | 1 | 1 | 4 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Progressive disease | 3 | 2 | 2 | 3 | 2 | 21 | 3 | 1 | 5
Not completed — Patient/Investigator request | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part A: Dose Escalation 600/5/NA: PXD101: 600 mg/m2 30-minute IV infusion every 24 hours for 5 days every 3 weeks (period of 3 weeks is one cycle) Carboplatin: AUC 5 administered 2-3 hours after PXD101 on Cycle Day 3 Paclitaxel: 0 mg/m2 administered 2-3 hours after PXD101 on Cycle Day 3
- Total: Total of all reporting groups
Arm/Group | Part A: Dose Escalation 600/5/NA | Part A: Dose Escalation 600/NA/175 | Part A: Dose Escalation 600/5/175 | Part A: Dose Escalation 800/5/175 | Part A: Dose Escalation 1000/5/175 | Part B: Ovarian Cancer MTD | Part C: 3 Hours Infusion, Solid Tumors Except Ovarian Cancer | Part C: 6 Hours Infusion Solid Tumors, Except Ovarian Cancer | Part D: Bladder Cancer MTD | Total
Number analyzed (Participants) | 5 | 5 | 3 | 4 | 6 | 35 | 4 | 3 | 15 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 3 | 4 | 6 | 22 | 4 | 3 | 8 | 59
  >=65 years | 0 | 1 | 0 | 0 | 0 | 13 | 0 | 0 | 7 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 0 | 3 | 35 | 3 | 1 | 4 | 52
  Male | 3 | 4 | 0 | 4 | 3 | 0 | 1 | 2 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerable Dose (MTD) Belinostat, Part A,
Description: To determine the maximum tolerated dose of belinostat (PXD101) in doses up to 1000 mg/m²/day administered in combination with standard doses of carboplatin (AUC of 5) and paclitaxel (175 mg/m2).
Time Frame: Cycle 1
Measure: Number; unit: mg/m2
Groups:
- Part A: Belinostat: Dose escalating up to 1000 mg/m2 days 1-5 in a 21 day cycle; IV Paclitaxel: administered in an intravenous infusion 2-3 hours after PXD101 infusion on day 3 of a 21 day cycle Carboplatin: administered in an intravenous infusion after paclitaxel on day 3 of a 21 day cycle
Arm/Group | Part A
Number analyzed (Participants) | 23
mg/m2 | 1000

2. Secondary Outcome: Best Overall Response (CR or PR)
Description: Best overall responses were assessed by RECIST (Response Evaluation Criteria in Solid Tumors) criteria. Clinical tumor evaluation will take place after each cycle. Formal radiological evaluation after every 2 cycles. If a response is noted, a follow-up radiographic assessment must be performed 4 weeks (+ 1 week) after the response is noted
Time Frame: Throughout study until PD (progressive disease) or lost to follow up
Population: Primary efficacy analysis population, includes all patients who have been enrolled into the study and received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Part A: Dose Escalation 600/5/NA | Part A: Dose Escalation 600/NA/175 | Part A: Dose Escalation 600/5/175 | Part A: Dose Escalation 800/5/175 | Part A: Dose Escalation 1000/5/175 | Part B: Ovarian Cancer MTD | Part C: 3 Hours Infusion, Solid Tumors Except Ovarian Cancer | Part C: 6 Hours Infusion Solid Tumors, Except Ovarian Cancer | Part D: Bladder Cancer MTD
Number analyzed (Participants) | 5 | 5 | 3 | 4 | 6 | 35 | 4 | 3 | 15
participants | 1 | 0 | 0 | 0 | 1 | 15 | 0 | 0 | 4

3. Secondary Outcome: To Determine the Pharmacodynamic Effects of Belinostat (in the Combination) on Histone Acetylation in Peripheral Blood Mononuclear Cells (Selected Sites)
Time Frame: Throughout the study
Population: Histone acetylase analysis was planned, but not successful due to technical issues with the method.
Arm/Group | Part A
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Progression
Description: Time to progression, defined as the interval between the first dates of treatment until the first notation of disease progression. RECIST criteria
Time Frame: Throughout study
Population: Per protocol Population, includes all patients who have received at least two cycles (complete treatment days, dose reductions per protocol allowed) of study treatment and who have also had at least one post-baseline tumor assessment. Not done for Part A.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Part C: 3-6 Hours Infusion, Solid Tumors Except Ovarian Cancer: PXD: 1000 mg/m² was administered as a 3-6 hour IV infusion every 24 hours for 5 days on Day 1-5 every 3 weeks Paclitaxel: 175 mg/m² IV administered 2-3 hours following the infusion of PXD101 on cycle Day 3 Carboplatin: AUC of 5 IV administered 2-3 hours following the infusion of PXD101 on cycle Day 3 (carboplatin after paclitaxel)
Arm/Group | Part B: Ovarian Cancer MTD | Part C: 3-6 Hours Infusion, Solid Tumors Except Ovarian Cancer | Part D: Bladder Cancer MTD
Number analyzed (Participants) | 30 | 6 | 14
days | 195 [165 to 225] | 150 [57 to NA] — Too few observations | 136 [123 to NA] — Too few observations

5. Secondary Outcome: Time to Response
Description: Time to response (RECIST) was assessed as the interval between the first dates of treatment until the first notation of response.
Time Frame: Throughout study
Population: Includes patients with response, i.e. 15 patients in Part B, 0 patients in Part C, and 4 patients in Part D. Not done for Part A.
Measure: Median (Full Range); unit: days
Arm/Group | Part B: Ovarian Cancer MTD | Part C: 3-6 Hours Infusion, Solid Tumors Except Ovarian Cancer | Part D: Bladder Cancer MTD
Number analyzed (Participants) | 15 | 0 | 4
days | NA [35 to NA] — Insufficient number of participants with events |  | NA [29 to NA] — Insufficient number of participants with events

6. Secondary Outcome: Duration of Response
Description: Defined as interval from the time criteria for CR or PR are met, until the first date that recurrent or progressive disease is objectively documented.
Time Frame: Throughout study
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Arm/Group | Part B: Ovarian Cancer MTD | Part C: 3-6 Hours Infusion, Solid Tumors Except Ovarian Cancer | Part D: Bladder Cancer MTD
Number analyzed (Participants) | 15 | 0 | 4
days | NA [79 to NA] — Insufficient number of participants with events |  | NA [56 to NA] — Insufficient number of participants with events

7. Secondary Outcome: Belinostat Cmax
Time Frame: Cycle 1 day 1: Pre-Infusion, 0 min, 5 min, 15 min, 30 min, 1 h, 2 h, 3 h, 3 h 15 min, 3 h 30 min, 4 h, 5 h, 6 h, 6 h 15 min, 6 h 30 min, 7h, 8h, 9h, 24h
Population: The Pharmacokinetic Analysis Subset consisted of 41 patients who enrolled in the study and provided a complete or partial set of pharmacokinetic parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Belinostat 600 mg/30 Minutes: PXD101: 600 mg/m2 30-minute IV infusion
- Belinostat 800 mg/30 Min: PXD101: 800 mg/m2 30-minute IV infusion
- Belinostat 1000 mg/30 Min: Belinostat 1000 mg/m2 30-minute IV infusion
- Belinostat 1000 mg/3-hours: Belinostat: 1000 mg/m² was administered as a 3 hour IV infusion every 24 hours
- Belinostat 1000 mg/6-hours: Belinostat 1000 mg/m² was administered as a 6-hour IV infusion every 24 hours
Arm/Group | Belinostat 600 mg/30 Minutes | Belinostat 800 mg/30 Min | Belinostat 1000 mg/30 Min | Belinostat 1000 mg/3-hours | Belinostat 1000 mg/6-hours
Number analyzed (Participants) | 12 | 4 | 18 | 4 | 3
ng/mL | 18592 (4390) | 22525 (6002) | 31517 (12684) | 8340 (635) | 2873 (210)

8. Secondary Outcome: Belinostat Mean t½
Time Frame: Cycle 1 Day 1: Cycle 1 day 1: Pre-Infusion, 0 min, 5 min, 15 min, 30 min, 1 h, 2 h, 3 h, 3 h 15 min, 3 h 30 min, 4 h, 5 h, 6 h, 6 h 15 min, 6 h 30 min, 7h, 8h, 9h, 24h
Population: The Pharmacokinetic Analysis Subset consisted of 39 patients who enrolled in the study and provided a complete or partial set of pharmacokinetic parameters
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Belinostat 600 mg/30 Minutes | Belinostat 800 mg/30 Min | Belinostat 1000 mg/30 Min | Belinostat 1000 mg/3-hours | Belinostat 1000 mg/6-hours
Number analyzed (Participants) | 11 | 4 | 18 | 4 | 2
hours | 1.41 (0.58) | 1.16 (0.133) | 0.898 (0.161) | 3.76 (2.9) | 1.9 (0.286)

9. Secondary Outcome: Belinostat AUC (0-infinity)
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Belinostat 600 mg/30 Minutes | Belinostat 800 mg/30 Min | Belinostat 1000 mg/30 Min | Belinostat 1000 mg/3-hours | Belinostat 1000 mg/6-hours
Number analyzed (Participants) | 11 | 4 | 18 | 4 | 2
ng*h/mL | 9116 (1670) | 11785 (2445) | 21057 (11034) | 31515 (3612) | 13107 (1004)

10. Primary Outcome: Dose Limiting Toxicities (DLT), Part A
Description: To determine the number of participants experiencing dose limiting toxicities of belinostat (PXD101) in doses up to 1000 mg/m²/day administered in combination with standard doses of carboplatin and paclitaxel or both.
Time Frame: Cycle 1
Measure: Number; unit: participants
Arm/Group | Part A
Number analyzed (Participants) | 23
participants | 0

ADVERSE EVENTS:
Groups:
- Part A: Dose Escalation (N=23); Part B: Ovarian Cancer MTD (N=35): PXD101: 1000 mg/m2 30-minute IV infusion every 24 hours for 5 days every 3 weeks (period of 3 weeks is one cycle) Carboplatin: AUC 5 administered 2-3 hours after PXD101 on Cycle Day 3 Paclitaxel: 175 mg/m2 administered 2-3 hours after PXD101 on Cycle Day 3
- Part C: 3-6 Hours Infusion (N=7): PXD: 1000 mg/m² was administered as a 3 or 6 hour IV infusion every 24 hours for 5 days on Day 1-5 every 3 weeks Paclitaxel: 175 mg/m² IV administered 2-3 hours following the infusion of PXD101 on cycle Day 3 Carboplatin: AUC of 5 IV administered 2-3 hours following the infusion of PXD101 on cycle Day 3 (carboplatin after paclitaxel)
- Part D: Bladder Cancer MTD (N=15): PXD101: 1000 mg/m² 30-minute IV infusion every 24 hours for 5 days on Day 1-5 every 3 weeks Carboplatin: AUC 5 IV, 2-3 hours following the infusion of PXD101 on Cycle Day 3 Paclitaxel: 175 mg/m² IV, 2-3 hours following the infusion of PXD101 on Cycle Day 3
Arm/Group | Part A: Dose Escalation (N=23) | Part B: Ovarian Cancer MTD (N=35) | Part C: 3-6 Hours Infusion (N=7) | Part D: Bladder Cancer MTD (N=15)
Serious Adverse Events (participants affected / at risk) | 17/23 | 19/35 | 7/7 | 7/15
Other Adverse Events (participants affected / at risk) | 23/23 | 35/35 | 7/7 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Dose Escalation (N=23) (N=23) | Part B: Ovarian Cancer MTD (N=35) (N=35) | Part C: 3-6 Hours Infusion (N=7) (N=7) | Part D: Bladder Cancer MTD (N=15) (N=15)
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Central Line Infection (Infections and infestations) | 2 | 1 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Disease Progression (General disorders) | 3 | 0 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 2
ECG Signs Of Myocardial Ischaemia (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT Corrected Interval Prolonged (Investigations) | 1 | 0 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 1 | 0 | 0 | 0
Thrombophlebitis Septic (Infections and infestations) | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhagic Disorder (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 2 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Drug Intolerance (General disorders) | 0 | 0 | 1 | 0
Enterococcal Infection (Infections and infestations) | 0 | 0 | 1 | 0
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal Stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection Enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram T Wave Inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenic Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral Motor Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureteric Haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vena Cava Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Dose Escalation (N=23) (N=23) | Part B: Ovarian Cancer MTD (N=35) (N=35) | Part C: 3-6 Hours Infusion (N=7) (N=7) | Part D: Bladder Cancer MTD (N=15) (N=15)
Nausea (Gastrointestinal disorders) | 16 | 34 | 7 | 11
Fatigue (General disorders) | 18 | 32 | 7 | 11
Oedema Peripheral (General disorders) | 4 | 9 | 1 | 4
Pyrexia (General disorders) | 4 | 6 | 7 | 5
Chills (General disorders) | 3 | 3 | 0 | 2
Disease progression (General disorders) | 3 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 5 | 0 | 2
Catheter Site Pain (General disorders) | 1 | 3 | 0 | 0
Mucosal Inflammation (General disorders) | 0 | 3 | 0 | 2
Chest Discomfort (General disorders) | 0 | 2 | 0 | 0
Face Oedema (General disorders) | 0 | 2 | 0 | 0
Localised Oedema (General disorders) | 0 | 2 | 0 | 0
Pain (General disorders) | 0 | 2 | 0 | 0
Drug intolerance (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 4
Catheter site phlebitis (General disorders) | 0 | 1 | 0 | 1
Injection site reaction (General disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 14 | 20 | 7 | 12
Vomiting (Gastrointestinal disorders) | 14 | 25 | 5 | 8
Diarrhoea (Gastrointestinal disorders) | 11 | 25 | 4 | 9
Abdominal pain (Gastrointestinal disorders) | 4 | 17 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 11 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 10 | 3 | 2
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 5 | 4
Flatulence (Gastrointestinal disorders) | 0 | 4 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 3 | 1
Small intestine obstruction (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Gastrooesophagela reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Lip blister (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Rectal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 14 | 24 | 6 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 15 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 16 | 2 | 5
Leukopenia (Blood and lymphatic system disorders) | 1 | 14 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 11 | 5 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 12 | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 9 | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 8 | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 10 | 25 | 6 | 10
Headache (Nervous system disorders) | 9 | 12 | 7 | 6
Dizziness (Nervous system disorders) | 6 | 15 | 4 | 1
Dysgeusia (Nervous system disorders) | 6 | 17 | 1 | 2
Paraesthesia (Nervous system disorders) | 2 | 1 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 3 | 1 | 0
Syncope (Nervous system disorders) | 0 | 3 | 0 | 1
Migraine (Nervous system disorders) | 0 | 2 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 3
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 3
Neurotoxicity (Nervous system disorders) | 0 | 1 | 0 | 2
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 26 | 6 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 6 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 8 | 3 | 5
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 11 | 5 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 10 | 3 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 12 | 15 | 7 | 4
Deep vein thrombosis (Vascular disorders) | 2 | 3 | 0 | 0
Hypertension (Vascular disorders) | 2 | 3 | 1 | 6
Hot flush (Vascular disorders) | 0 | 4 | 0 | 0
Hypotension (Vascular disorders) | 0 | 4 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 2 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 1 | 0 | 2
Diastolic hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 10 | 12 | 7 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 11 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 9 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 8 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 7 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 7 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 5 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 9 | 0 | 5
Central line infection (Infections and infestations) | 2 | 1 | 0 | 2
Oral candidiasis (Infections and infestations) | 2 | 3 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 5 | 2 | 0
Candidiasis (Infections and infestations) | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 2 | 0
Bacteriaemia (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 3 | 1 | 2 | 0
Blood potassium decreased (Investigations) | 2 | 1 | 1 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 | 1 | 0 | 0
White blood cell count increased (Investigations) | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 7 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 7 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 6 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 0 | 0
Blood glucose increased (Investigations) | 0 | 2 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 2 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 11 | 4 | 1
Anxiety (Psychiatric disorders) | 2 | 5 | 0 | 0
Depression (Psychiatric disorders) | 2 | 4 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 3 | 3 | 0 | 1
Palpitations (Cardiac disorders) | 2 | 3 | 4 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 2 | 8 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1
Bladder pain (Renal and urinary disorders) | 2 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 5 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 4 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 3 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 2 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 4 | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureteric haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urethral haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 8 | 3 | 4
Hypersensitivity (Immune system disorders) | 1 | 2 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 3 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 3 | 0 | 0
Genital pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 1 | 0 | 2 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ureteric diversion operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less